CLINICAL TRIAL: NCT04817124
Title: Feasibility of Cognitive Training in Combination With Transcranial Direct Current Stimulation in a Home-based Context
Brief Title: Cognitive Training Combined With Transcranial Direct Current Stimulation in Older Adults in a Home-based Context
Acronym: TrainStim4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TrainStim4
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Aging
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation group (Experimental): Anodal tDCS+ intensive cognitive Training
  Interventions: Device: Anodal tDCS; Behavioral: Intensive cognitive training
- sham group (Sham Comparator): Sham tDCS + intensive cognitive Training
  Interventions: Behavioral: Intensive cognitive training; Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — Anodal transcranial direct current stimulation (tDCS), 6 sessions with 20 minutes stimulation each (1,5 mA).
  Arms: stimulation group
Behavioral: Intensive cognitive training — Intensive cognitive training of a letter memory updating task, 6 sessions for approximately 20 min
Device: Sham tDCS — Sham transcranial direct current stimulation (tDCS), 6 sessions with 30 sec stimulation each (1,5 mA) to ensure blinding of participants.
  Arms: sham group

SUMMARY:
The aim of this study is to investigate whether a tDCS-accompanied intensive cognitive training is feasible as a home-based intervention.

DETAILED DESCRIPTION:
The goal of the present study is to assess feasibility (primary) and cognitive training and transfer effects of a home-based multi-session cognitive training combined with transcranial direct current stimulation (tDCS). tDCS, particularly in combination with cognitive training, represents a promising approach to counteract cognitive decline and restore impaired functions. However, combined interventions of cognitive training and tDCS involve frequent visits to the facility, which leads to the need of space, time and personnel, and imposes strains on the participants. This study will elucidate the feasibility of tDCS and cognitive training in a home-based context. Healthy older adults will participate in a two-week cognitive training with concurrent online tDCS application in their own homes. Feasibility, as well as cognitive performance will be examined before, during and after the intervention. In order to draw conclusions about the effect of tDCS in addition to cognitive training, a control group, receiving sham stimulation during training, will be assessed. A Follow-up session to assess long-term effects is planned four weeks after the post assessment. We hypothesize that with appropriate training of the participants and close supervision the use of combined tDCS and cognitive training in an ecologically valid environment by the participants themselves is feasible. In addition, we hypothesize this protocol will lead to improved performance on the trained tasks in both experimental groups. We expect increased performance on transfer tasks and long-term maintenance of the effects after anodal compared to sham stimulation. A successful implementation of the intervention in the home-based setting will contribute to the development of home-based tDCS as a widely available therapy option in clinical populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 60 - 80 years
2. Right handedness

Exclusion Criteria:

1. Neurodegenerative neurological illnesses, epilepsy or history of seizures
2. Severe and untreated medical conditions that preclude participation in the training, as determined by responsible physician
3. History of severe alcoholism or use of drugs
4. Severe psychiatric disorders such as depression (if not in remission) or psychosis
5. Contraindication to tDCS application

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting the intervention in a home-based context | 2 weeks
  Feasibility of home-based tDCS as operationalized by at least 2/3 (out of 6 planned sessions) successfully performed interventional sessions per participant. A session is regarded as successful if it is marked as completed in the stimulation system.

SECONDARY OUTCOMES:
Feasibility (questionnaire) | 2 weeks
  Self-rate questionnaire of participant satisfaction, independence and self-confidence in the handling of the devices and program (cf. Cha at el., 2016) after training period (anodal condition versus sham)
Working memory performance at post-assessment | 2 weeks
  Performance in a near transfer task (n-back) under anodal tDCS compared to sham condition; operationalized by % correct responses in the n-back task
Working memory performance at follow-up assessment | 4 weeks after intervention
  Performance in a near transfer task (n-back) under anodal tDCS compared to sham condition; operationalized by % correct responses in the n-back task
Working memory training performance (Letter Updating Task) at post-assessment | 2 weeks
  Performance in primary memory training task (Letter Updating Task) at post-assessment, operationalized by number of correctly recalled lists in the letter updating task
Working memory training performance (Letter Updating Task) at follow-up assessment | 4 weeks after intervention
  Performance in primary memory training task (Letter Updating Task) at follow-up assessment, operationalized by number of correctly recalled lists in the letter updating task

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof., Study Director — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Thams F, Rocke M, Malinowski R, Nowak R, Grittner U, Antonenko D, Floel A. Feasibility of Cognitive Training in Combination With Transcranial Direct Current Stimulation in a Home-Based Context (TrainStim-Home): study protocol for a randomised controlled trial. BMJ Open. 2022 Jun 10;12(6):e059943. doi: 10.1136/bmjopen-2021-059943. PMID 35688585

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT04817124/SAP_000.pdf